CLINICAL TRIAL: NCT04440579
Title: Utilization of Percutaneous Tibial Nerve Stimulation During Office-Based Cystoscopy: A Pilot Study
Brief Title: Utilization of PTNS During Office-Based Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Holzbeierlein, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 145954
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cystoscopy
Keywords: Cystoscopy; Urology

STUDY DESIGN:
Masking Description: This study will be a double-blind, randomized control trial, with one additional unblinded arm. The two blinded arms will be PTNS and sham PTNS, with the additional unblinded arm being standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Cystoscopy (Active Comparator): Patients will undergo a standard of care cystoscopy
  Interventions: Procedure: Standard Cystoscopy
- PTNS and Cystoscopy (Experimental): Patients will undergo PTNS while undergoing cystoscopy
  Interventions: Procedure: Percutaneous Tibial Nerve Stimulation (PTNS); Procedure: Standard Cystoscopy
- Sham PTN and Cystoscopy (Sham Comparator): Patients will undergo a sham PTNS procedure while undergoing cystoscopy
  Interventions: Procedure: Sham Percutaneous Tibial Nerve Stimulation (PTNS); Procedure: Standard Cystoscopy

INTERVENTIONS:
Procedure: Percutaneous Tibial Nerve Stimulation (PTNS) — PTNS is neuromodulation that uses electricity to stimulate the nervous system, specifically the posterior tibial nerve, and is minimally invasive.
  Arms: PTNS and Cystoscopy
Procedure: Sham Percutaneous Tibial Nerve Stimulation (PTNS) — Patients will be connected to the PTNS device but the device will remain off for the entirety of the procedure
  Arms: Sham PTN and Cystoscopy
Procedure: Standard Cystoscopy — Patient will undergo standard cystoscopy

SUMMARY:
This study will be a double-blind, randomized control trial, with one additional unblinded arm. This study has been designed to identify a means of improving quality of life for patients requiring in-office cystoscopy. Percutaneous tibial nerve stimulation (PTNS) has been shown to improve quality of life and symptom control in multiple urological conditions based on shared neuroanatomical structures between the genitourinary system and the tibial nerve The goal of this project is to demonstrate the efficacy and safety of PTNS in minimizing patient discomfort during cystoscopy to develop a larger randomized control trial in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients undergoing routine office-based cystoscopy by a urology provider

Exclusion Criteria:

* Patients for whom ancillary procedures are performed during cystoscopy, including ureteral stent removal, bladder stone removal, biopsy, or fulguration
* Patients undergoing cystoscopy due to concern for urologic injury
* Patients undergoing cystoscopy due to concern for prosthetic abnormality, including erosion or malposition
* Patients who perform clean intermittent catheterization
* Patients with pre-existing neurological pathology, including but not limited to multiple sclerosis, spinal cord injury, Parkinson's disease, or peripheral neuropathy of any etiology
* Patients having undergone prior non-endoscopic prostatectomy (radical prostatectomy, simple prostatectomy)
* Patients with a history of interstitial cystitis/chronic pelvic pain
* Patients who have taken an analgesic (excluding 81mg aspirin) in the past 12 hours
* Patients with a history of urethral stricture disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Patient Discomfort | One year
  To assess the ability of percutaneous tibial nerve stimulation to improve patient discomfort during routine office-based cystoscopy based on a 10-point visual analogue scale (VAS) by comparing median and interquartile ranges between groups. A score of 0 will indicate no pain whereas a score of 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Safety of PTNS: adverse events | One year
  To determine the safety of PTNS for use in the setting of routine office-based cystoscopy based on rate of adverse events as defined by the Clavien-Dindo classification system

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Holzbeierlein, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No